CLINICAL TRIAL: NCT05780879
Title: A Proof of Concept Pilot Study of the Addition of Venetoclax to Standard Remission Induction Chemotherapy Fludarabine or Cladrabine, Cytarabine, and Granulocyte Colony Stimulating Factor (G-CSF) (FLAG or CLAG) for Frontline Therapy of Secondary Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2021.145; HUM00227799 (Other: University of Michigan)
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Secondary Acute Myeloid Leukemia
MeSH Terms: interventions — venetoclax; CLAG protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax + FLAG or CLAG induction chemotherapy (Experimental): Induction chemotherapy with FLAG starting on day 1 and venetoclax given on days 3-16. The G-CSF component of FLAG will continue until count recovery (ANC at least > 1000). FLAG dosing will be standard and uniform for all patients and venetoclax dosing will be determined according to institutional guidelines based on the prophylactic antifungal therapy chosen for use during induction therapy. Given the national shortage of Fludarabine, Cladrabine (5mg/m2/day IV over 2 hours) has been substituted (CLAG) with similar toxicity profile.
  Interventions: Drug: Venetoclax; Drug: FLAG or CLAG Protocol

INTERVENTIONS:
Drug: Venetoclax — Venetoclax administered orally once daily on days 3-16.
Drug: FLAG or CLAG Protocol — FLAG consists of daily infusions of Fludarabine (30mg/m2/day over 30 minutes) and Ara-C (2g/m2/day over 4 hours) for 5 days with daily subcutaneous injections of G-CSF until count recovery. Tbo-filgrastim will be administered as follows: WBC count >50,000 - 5mcg/kg; WBC count <50,000 - hold Tbo-filgrastim. Given the national shortage of Fludarabine, Cladrabine (5mg/m2/day IV over 2 hours) has been substituted (CLAG) with similar toxicity profile.

SUMMARY:
The primary purpose of this study is to determine complete remission rate of a novel combination induction chemotherapy treatment based upon 20 patients with newly diagnosed secondary AML.

ELIGIBILITY:
Inclusion Criteria:

* Patients have an established, pathologically confirmed diagnosis of newly diagnosed secondary acute myeloid leukemia (sAML) as defined by the 2016 World Health Organization criteria. Secondary AML includes:

  * AML arising after an antecedent hematologic neoplasm including aplastic anemia (AA), myelodysplastic syndrome (MDS), myeloproliferative neoplasms (MPNs), and overlap syndromes (MDS/MPN)
  * AML with MDS defining cytogenetic changes as defined in Vardiman et al. Blood 2009 114 (5): 937-951 - Table 6. Please see appendix 14.6 for full table.
  * Therapy-related AML
* Patients must not have received prior treatment for the diagnosis of secondary acute myeloid leukemia, with the exception of hydroxyurea and/or leukopheresis which are permitted until day 1 of study participation. Prior treatment for a diagnosis of MDS, MPN, or MDS/MPN overlap syndrome is allowed.
* Patients ≥ 18 years of age.
* ECOG PS ≤ 2
* Patient has ability to understand and the willingness to sign a written informed consent.
* Adequate organ function as defined by:

  * serum creatinine level ≤ 2.0 mg/dL or a CrCl ≥ 30 ml/min (Cockcroft-Gault equation using actual body weight)
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤ 3 times the institutional upper limit of normal (ULN) unless considered due to leukemic involvement
  * total bilirubin level ≤1.5 times the institutional upper limits of normal (ULN) (unless secondary to Gilbert syndrome, hemolysis, or suspected leukemic involvement).
* Patients must be non-fertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception associated with a low failure rate during and for at least 6 months after completion of study therapy.
* Patients must be able to comply with the requirements for the entire duration of the study.

Exclusion Criteria:

* Diagnosed with acute promyelocytic leukemia (acute leukemia with recurrent genetic abnormalities - APL with t(15;17)(q22;q12);PML-RARA).
* Diagnosed with myeloid blast phase of chronic myeloid leukemia.
* Diagnosed with isolated extramedullary AML
* Diagnosed with acute leukemia of ambiguous lineage, acute biphenotypic or acute bilineal acute leukemia per the 2016 World Health Organization classification system.
* Patients with a white blood cell count (WBC) >50,000 at the time of initiation of therapy will be excluded. Patients can consent and screen with a WBC > 50,000 but will require cytoreduction (hydrea or leukopheresis) prior to day 1 of therapy.
* Receiving antileukemic therapy other than hydroxyurea. Patients may have received therapy with a hypomethylating agent (azacitidine or decitabine) for a prior diagnosis of myelodysplastic syndrome (MDS) or chemotherapy for a prior diagnosis of a myeloproliferative neoplasm or an MDS/MPN overlap syndrome. Likewise, patients may have received chemotherapy for a prior non-leukemic oncologic malignancy.
* Any prior therapy with a Bcl-2 antagonist.
* Any known allergy to the chemotherapeutic agents being investigated including fludarabine,cladribine, cytarabine, G-CSF and venetoclax.
* Clinical signs of active leptomeningeal leukemia or biopsy proven active leptomeingeal leukemia. A clinical history of previously treated leptomeningeal process is not exclusionary.
* Patients with known history of HIV, Hepatitis B, or Hepatitis C with the exception of those with an undetectable viral load within 3 months of screening. (Hepatitis B or C testing is not required). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate.
* Having an active second malignancy requiring treatment--other than AML--within 3 months prior to the start of treatment, with the exception of basal cell carcinoma or squamous cell carcinoma of the skin, colon polyp, carcinoma in situ of the cervix, or DCIS/LCIS of the breast.
* Having an active uncontrolled infection (viral, bacterial or fungal), any other concurrent disease, or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator.
* Pregnant women or women who are breastfeeding. Women must be willing to not breast feed up until 30 days following the end of trial therapy.
* Men or women of childbearing potential must be willing to practice an effective method of birth control during treatment and up until 6 months following the end of trial therapy.
* Having received any live vaccines within 28 days prior to first study drug administration.
* Patient has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
* Patient has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Patient has a cardiovascular disability status of New York Heart Association Class > 2.
* Patient has a chronic respiratory disease that requires continuous supplemental oxygen.
* Patient has a malabsorption syndrome or other condition that precludes enteral route of administration of medications.
* Female subject that has positive results for a screening pregnancy test.

  * Women of childbearing potential are defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception defined as:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    * Male sterilization (at least six months prior to enrolling). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
    * Use of a combination of any two of the following:

      * Use of oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormonal vaginal ring or transdermal hormone contraception.
      * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/cream/vaginal suppository.
  * Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to enrolling. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
  * If a study patient becomes pregnant or suspects being pregnant during the study or within 30 days after the final dose of trial therapy, the Study Doctor needs to be informed immediately.
* Malabsorption syndrome or other condition that would interfere with enteral absorption or an inability to take oral medications as prescribed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Morphologic complete remission (CR) | up to 43 days (+/- 2 days)
  If at least 12/20 (60%) of patients achieve a CR (based upon a bone marrow aspiration, biopsy, and peripheral blood studies according to the International Working Group criteria for AML), the combination treatment will be considered successful. If the true CR rate is 40%, then the trial will be considered successful with probability 0.06 (type I error). Conversely, if the true CR rate is 70%, then the trial will be considered successful with probability 0.89 (power).
Percentage of patients who develop drug-related non-hematologic grade 3 or higher toxicity | 30 days post study treatment start
  Percent of patients who develop drug-related non-hematologic grade 3 or higher toxicities within 30 days after study treatment initiation (excluding nausea and vomiting or electrolyte abnormalities that are corrected with standard clinical care).
Number of patients who develop drug-related non-hematologic grade 3 or higher toxicity | 30 days post study treatment start
  Number of patients who develop drug-related non-hematologic grade 3 or higher toxicities within 30 days after study treatment initiation (excluding nausea and vomiting or electrolyte abnormalities that are corrected with standard clinical care).
Bone marrow aplasia | up to 43 days (+/- 2 days)
  Defined as a bone marrow biopsy with an overall cellularity of < 5% with no evidence of leukemia as well as an ANC <0.5 and a platelet count of < 10 requiring transfusion support.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 28 days (+/- 7 days) days post remission marrow collection
  {Percentage of patients?} with complete remission (CR), complete remission with incomplete count recovery (CRi), morphologic leukemia free state rate (MLFS), and partial response rate (PR) per AML Response Criteria.
Progression-free survival (PFS) | 6 months and 1 year following the conclusion of study enrollment
  PFS defined as the time between first dose of study treatment to the event of disease progression or death; analyzed using Kaplan Meier methods.
Overall survival (OS) | 6 months and 1 year following the conclusion of study enrollment
  OS defined as the time from start of treatment to death; analyzed using Kaplan Meier methods.
Event free survival (EFS) | 6 months and 1 year following the conclusion of study enrollment
  EFS defined as the time from start of treatment to resistant leukemia, relapsed leukemia, second malignancy, or death; analyzed using Kaplan Meier methods.
Mortality rate | 30 days post study treatment start
  Defined as whether the patient was alive 30 days post-study treatment start (died/not died).
Allogeneic transplantation | 1 year after study entry
  Defined as the total number of patients requiring allogeneic transplantation after protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Bixby, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No